CLINICAL TRIAL: NCT04415437
Title: Self-Stigma of Mental and Physical Health: Developing and Validation of a Universal Self-Stigma Scale (USSS)
Brief Title: Self-Stigma of Mental and Physical Health
Status: Completed | Type: Observational
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-53k
Record Dates: First submitted 2020-05-06; First posted 2020-06-04 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Mental Disorder; Organic Disease
Keywords: Self-Stigma; Mental Health; Physical Health; Questionnaire
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy: Healthy participants
- mentally ill: Participants with mental disorders
- physically ill: Participants with organic disease
- mentally and physically ill: Participants with mental disorders and organic disease

SUMMARY:
People with mental disorders often suffer from self-stigmatization. Self-stigma is associated with several negative outcomes such as low quality of life, lower rates of help-seeking as well as poorer treatment adherence. However, a lot of questionnaires only focus on specific mental disorders. There is no valid measurement which can be used for all kinds of mental disorders.

Furthermore, much less is known about self-stigma in people with organic diseases. Only little attention has been given to those who may experience self-stigma because of their physical condition. A main reason for this may be the lack of a valid measurement of self-stigma among people with physical health issues.

Therefore, the aim of this study is to develop and validate a self-report scale which is capable to do both - measuring self-stigma among people with all mental disorders and among people with physical health issues.

DETAILED DESCRIPTION:
Items are derived from the Stereotype Content Model (SCM) and the Behaviors from Intergroup Affect and Stereotypes (BIAS) Map. Psychometric evaluation includes testing the reliability (intern consistency, test-retest reliability) and validity (exploratory and confirmatory factor analysis, construct validity incl. convergent and discriminant validity, criterion-related validity).

Participants take part in an online survey. They answer general questions about their mental and physical health condition and complete measurements of quality of life, mental health, depression, public stigma, expected stigma, self-stigma, intention to seek help and actual help seeking (behavior).

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age: 18
* Fluent in German Language

Exclusion Criteria:

* Acute psychosis
* Suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random sample including students, outpatients, inpatients
Sampling Method: Non-Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Development of the Universal Self-Stigma Scale (USSS) | Baseline
  Questionnaire is based on the Stereotype Content Model (Fiske et al., 2002) and BIAS-Map (Cuddy et al., 2007) and includes three components: stereotype (warmth, competence [lower scores indicate higher self-stigma]), prejudice (emotions, e.g. contempt, pity, anger, shame [higher scores indicate higher self-stigma]), discrimination (active/passive self-harm [higher scores indicate higher self-stigma]). Each item is rated on a 7-point Likert scale.
  Item selection via qualitative and statistical methods, e.g. item difficulty index, item discrimination index, exploratory factor analysis (EFA).
Universal Self-Stigma Scale (USSS): Validity | Baseline
  Validation process includes confirmatory factor analysis (CFA) to test the statistical model fit with goodness of fit indices. Convergent validity is tested with another measurement for self-stigma (ISMI) using Pearson correlations [higher correlations indicate better convergent validity]. Discriminant validity is tested with Beck Depression Inventory-II (BDI-II) and public stigma [lower correlations indicate better discriminant validity], criterion validity with actual help seeking behavior and health related quality of life (12-Item Short-Form Health Survey, SF-12) using Pearson correlations as well [higher correlations indicate better criterion validity].
Universal Self-Stigma Scale (USSS): Internal consistency | Baseline
  Internal consistency is tested with Cronbach's Alpha (0-1; higher scores indicate better internal consistency)
Change on Universal Self-Stigma Scale (USSS): Test-Retest Reliability | Baseline and 4 weeks
  Test-Retest Reliability (Pearson Correlation, 0-1; higher scores indicate better reliability)

SECONDARY OUTCOMES:
Intention to Seek Help | Baseline
  Questionaire (e.g. Yu et al., 2015) to describe the intention to seek help because of severe psychological or mental health problems as well as physical health problems (e.g. "If you had severe mental health problems, would you seek help from professional sources for them?", scores from 1 [definitely yes] to 4 [definitely no]; lower scores indicate higher intentions to seek help). Reasons for not seeking help because of psychological health problems (e.g. "I want to solve problems by myself.") are assessed by binary items (yes, no).
Actual Help Seeking Behavior | Baseline and 4 weeks
  8 Items to assess actual help seeking behavior. It is asked if participants have ever sought services from any professional and if they have been in therapy or received medical treatment because of psychological or physical health problems. As well as if they are using any of these services currently. Items are binary (yes, no).
12-Item Short-Form Health Survey (SF-12) | Baseline
  Self-report measure of health related quality of life; norm-based scores (M=50, SD=10) for Physical Component Summary (PCS) and Mental Component Summary (MCS), higher score indicates better health state
Patient Health Questionnaire (PHQ) | Baseline
  Self-report inventory used to screen for mental health disorders (depression, anxiety, alcohol, eating, somatoform disorders), including severity scores for depressive symptoms (0-29), anxiety symptoms (0-21) and somatic symptoms (0-30), where higher scores indicate more serve symptoms
Beck Depression Inventory-II (BDI-II) | Baseline
  Self-report measure of depressed mood; higher total scores indicate more servere symptoms; total score (0-63); cut-offs for interpretation 0-13 (minimal depression), 14-19 (mild depression), 20-28 (moderate depression), 29-63 (severe depression)
Public Stigma | Baseline
  Measuring public stigma including stereotype (cognition - warmth, competence), prejudice (emotions - pity, envy, contempt, admiration) and discrimination (behavior - active/passive harm) with 19 items based on Stereotype Content Model (Fiske et al., 2002) and BIAS Map (Cuddy et al., 2007) toward people with mental or physical health problems.
  (e.g. "How often do you think people in general tend to feel the following emotions toward people with a mental disorder? [pity, contempt, envy, admiration]")
Expected Stigma | Baseline and 4 weeks
  Expectation to be stigmatized because of one's own mental and physical health condition.
  (e.g. "Do you expect that other people think badly of you because of your health condition?")

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided